CLINICAL TRIAL: NCT02306395
Title: Endometrial Local Injury of Frozen Cycle to Improve the Outcome of Embryo Transfer of Repeated Implantation Failure.
Brief Title: Endometrial Local Injury to Improve the Outcome of Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY-2014
Record Dates: First submitted 2014-11-22; First posted 2014-12-03 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Female Infertility Due to Nonimplantation of Ovum
Keywords: endometrial local injury; repeated implatation failure; embyo transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial local injury (Experimental): Endometrial local injury is carried in the first 3-5 days after menstrual period at the same time of hysteroscopy.
  Interventions: Procedure: Endometrial local injury
- The blank group (No Intervention): Any processing does not carry on the endometrium in the first 3-5 days after menstrual period except hysteroscopy.

INTERVENTIONS:
Procedure: Endometrial local injury — The way of intervention is to scratch the uterine cavity two cycles by a small spatula in the first 3-5 days after menstrual period.
  Arms: Endometrial local injury

SUMMARY:
The purpose of this study is to determine whether edometrial local injury improves the outcome of embryo transfer,and to find out more evidence about the time of trauma,the way of intervention,and the possible mechanism.

DETAILED DESCRIPTION:
It is important to evaluate the efficacy of endometrial local injury in assisted reproductive technology(ART),especially on the patients of recurrent implantation failure. Although most trials proved the effectiveness of the intervention of local injury, the subjects of these trials are rarely the patients of repeated implantation failure(RIF). Moreover, the mechanism of endometrial injury is not clear.Our trial may provide further basis for this purpose by comparing to the quality of endometrium in two-dimensional ultrasound.If the technique demonstrates efficacy, it would help the patients with RIF caused by poor conditions of endometrium to deal with the problem of infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women with RIF(≥2) of embyo transfer and uneven echo of endometrium on HCG day(12-14 days)
* Without operation history of uterine cavity in the previous three months
* Who agree to join in the study

Exclusion Criteria:

* Women more than 40 years or less than 20 years
* With infectious diseases or endocrine diseases
* Who refuse to participate in the experiment

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
implantation rate | 3 months after intervention
  When serum HCG is continuously more than 100mIU/ml and gestational sac is detected by ultrasound,it is considered as implantation.

SECONDARY OUTCOMES:
the change of three-dimensional ultrasound of uterine cavity before and after intervention | in implantation window period(12-14 days)
  including endometrial thickness, echo, blood flow and uterine cavity volume, uterine vascularization index, flow index.
clinical pregnancy rate | an expected average of 7 week after pregnancy
  The standards is to detect fetal heart beat by ultrasound.
live birth rate | follow-up for one year after pregnancy
  The statistical ratio of live birth rate in two groups
the rate of birth defects | follow-up for one year after pregnancy
  calculate the rate of birth defects in two groups
the expression changes of endometrial inflammatory factors | endometrial sampling after local injury ,in the first 3-5 days after menstrual period
  Detection of inflammatory factors, such as LIF,MIP-1.
  ---------------------------
infection rate | one week after intervention
  detection of infection by serum test

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Wang, Dr, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Department of Obstetrics and Gynecology, Navy General Hospital., Beijing, Beijing Municipality, China

REFERENCES:
- [Background] El-Toukhy T, Sunkara S, Khalaf Y. Local endometrial injury and IVF outcome: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Oct;25(4):345-54. doi: 10.1016/j.rbmo.2012.06.012. Epub 2012 Jun 26. PMID 22885017
- [Background] Potdar N, Gelbaya T, Nardo LG. Endometrial injury to overcome recurrent embryo implantation failure: a systematic review and meta-analysis. Reprod Biomed Online. 2012 Dec;25(6):561-71. doi: 10.1016/j.rbmo.2012.08.005. Epub 2012 Sep 12. PMID 23063812
- [Background] Zhou L, Li R, Wang R, Huang HX, Zhong K. Local injury to the endometrium in controlled ovarian hyperstimulation cycles improves implantation rates. Fertil Steril. 2008 May;89(5):1166-1176. doi: 10.1016/j.fertnstert.2007.05.064. Epub 2007 Aug 6. PMID 17681303
- [Result] Finn CA, Martin L. Endocrine control of the timing of endometrial sensitivity to a decidual stimulus. Biol Reprod. 1972 Aug;7(1):82-6. doi: 10.1093/biolreprod/7.1.82. No abstract available. PMID 5050152
- [Result] Narvekar SA, Gupta N, Shetty N, Kottur A, Srinivas M, Rao KA. Does local endometrial injury in the nontransfer cycle improve the IVF-ET outcome in the subsequent cycle in patients with previous unsuccessful IVF? A randomized controlled pilot study. J Hum Reprod Sci. 2010 Jan;3(1):15-9. doi: 10.4103/0974-1208.63116. PMID 20607003
- [Result] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877
- [Result] Karimzade MA, Oskouian H, Ahmadi S, Oskouian L. Local injury to the endometrium on the day of oocyte retrieval has a negative impact on implantation in assisted reproductive cycles: a randomized controlled trial. Arch Gynecol Obstet. 2010 Mar;281(3):499-503. doi: 10.1007/s00404-009-1166-1. Epub 2009 Jul 1. PMID 19568761
- [Result] Baum M, Yerushalmi GM, Maman E, Kedem A, Machtinger R, Hourvitz A, Dor J. Does local injury to the endometrium before IVF cycle really affect treatment outcome? Results of a randomized placebo controlled trial. Gynecol Endocrinol. 2012 Dec;28(12):933-6. doi: 10.3109/09513590.2011.650750. Epub 2012 Sep 3. PMID 22943664
- [Result] Parsanezhad ME, Dadras N, Maharlouei N, Neghahban L, Keramati P, Amini M. Pregnancy rate after endometrial injury in couples with unexplained infertility: A randomized clinical trial. Iran J Reprod Med. 2013 Nov;11(11):869-74. PMID 24639710
- [Result] Gnainsky Y, Granot I, Aldo PB, Barash A, Or Y, Schechtman E, Mor G, Dekel N. Local injury of the endometrium induces an inflammatory response that promotes successful implantation. Fertil Steril. 2010 Nov;94(6):2030-6. doi: 10.1016/j.fertnstert.2010.02.022. Epub 2010 Mar 24. PMID 20338560